CLINICAL TRIAL: NCT05870020
Title: Validation of a Quality of Life Assessment Tool in Generalized Dystonodyskinetic Syndromes Treated With Continuous Electrical Neuromodulation (CEN): The "Dystono-dyskinetic BrethoméSanrey Quality of Life" Scale (DBS-QoLs)
Brief Title: Validation of a Quality of Life Assessment Tool in Adult Generalized Dystonodyskinetic Syndromes Treated by Continuous Electrical Neuromodulation
Acronym: DBS-QoLs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL22_0228
Record Dates: First submitted 2023-04-06; First posted 2023-05-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Dystono-dyskinetic Syndromes
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with dystono-diskinetic syndrome treated by depp brain stimulation in the unit. (Experimental)
  Interventions: Other: Questionnaire (DBS-QoLs)

INTERVENTIONS:
Other: Questionnaire (DBS-QoLs) — The DBS-QoLs questionnaire will be sent to the patients for answer:
  The questonnaire will be sent at :
  * the inclusion
  * 15 days after the inclusion
  * 1 year after the inclusion

SUMMARY:
In spite of a growing interest in the evaluation of health-related quality of life in movement's disorders management, there is no tool specifically dedicated to dystonia and related syndromes that measures both the objective severity of the handicap and the patient's feelings about the surgical treatment in terms of subjective improvement. We have been working for several years at the bedside of patients operated on in the " pathologies cérébrales résistantes " Unit on the development of a related questionnaire to assess both the motor severity and the patients' feelings about the evolution of their disease under Deep Brain Stimulation (DBS).

The self-questionnaire designed would allow to a certain extent to get away from the two gold standards currently used in the field, i.e. the Burke, Fahn & Marsden Dystonia Rating Scale (BFMDRS) and the SF-36, thus facilitating the evaluation and allowing a homogenization of the practices for the different implanting centers on the french territory.

DETAILED DESCRIPTION:
The construction of the tool in its particular design, including various targeted modules, stems from an experience of more than ten years acquired with patients treated by deep brain stimulation in the unit. The self-questionnaire thus obtained will be sent to 146 patients with generalized dystonodyskinetic syndrome, operated and followed in the unit, and submitted to various statistical analyses. The scores of the identified dimensions will be compared with the etiology of the abnormal movements (primary vs. secondary) as well as with the results obtained with the two scales currently used to evaluate abnormal movements (BFMDRS) and/or quality of life (SF-36) and finally with the patients' mood during their follow-up (BDI, STAI). Tolerance to surgery will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adulte between 18 an 80 years
* Patient with a generalized dystono-dyskinetic syndrome treated by Electrical Neuromodulation Continue and follow-up in the unit
* Subject affiliated to the French social security system

Exclusion Criteria:

* non-French speaker
* patients who are physically unable to answer the questionnaire and who have no trusted person to help
* severe cognitive impairment (MoCA <10, MDRS <123, PM-38 <70)
* lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ability to perform different activities assessed by DBS-QOLs | 1 year
  Ability to perform different activities assessed by the Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale (DBS-QOLs) with the evaluation of the ability to perform different activities (from impossible to autonomous) and then to estimate the evolution of this ability since the intervention (worsening, no change, improvement)
Psycho-social assessment by DBS-QOLs | 1 year
  Psychosocial assessment by the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) with yes/no/partially questions related to the emotional and psychological perception of patients and then to estimate the evolution of this thought since the intervention (worsening, no change, improvement)
Intervention's assessment by DBS-QOLs | 1 year
  Intervention's assessment by "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) with yes/no question related to the intervention.
Life's Quality assessment by DBS-QOLs | 1 year
  Life's Quality assessment by "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) with squales from 0 (worst case) to 10 (best case).

SECONDARY OUTCOMES:
External validity of the DBS-QOLs compared to the BFMDRS for the functional subscale | 1 year
  Correlation between the "Functional" subscale of the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) and the total score obtained on the Functional dimension (Mobility + Activity of Daily Living) of the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs).
External validity of the DBS-QOLs compared to the Beck Depression Inventory score for Thumia | 1 year
  Correlation of the Thumia score assessed by the Beck Depression Inventory score & the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) through the answer the the emotional and psychological perception of patients which have 12 items (Impossible, third person help, technology help, autonomous)
External validity of the DBS-QOLs compared to the SF-36 for Life's quality | 1 year
  Comparison of the Life's quality assessed by the Short Form (36) Health Survey (SF-36) and by the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) with different yes/no question
External validity of the reproducibility of the DBS-QOLs compared to the BFMDRS | 1 year
  Comparison of the sentivity to change between the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) and the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) through the evolution of the answer of DBS-QoLs and BFMDRS during the following of the patient.
External validity according to different clinical criteria or scales : sensitivity to change | 1 year
  Sensitivity to change (assessment of changes during follow-up by the BFMDRS).
Assessment of the correlation between the functional fain & the benefit felt by the patient with the DBS-QOLs | 1 year
  Assessment of the correlation between the measure of benefit in terms of functional gain and the benefit experienced by the patient with all the answer of all module in "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs).
Assessment of the tolerance to surgery by the DBS-QOLs | 1 year
  Assessment of the tolerance to surgery through the "surgical" module of the "Dystono-dyskinetic Brethomé-Sanrey Quality of Life scale" (DBS-QOLs) which is composed of yes/no questions.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, Hérault, France